CLINICAL TRIAL: NCT01502904
Title: Neointimal Coverage After Implantation of Biolimus Eluting Stent With Biodegradable Polymer: Optical Coherence Tomographic Assessment According to the Treatment of Dyslipidemia and Hypertension and the Types of Implanted Drug-eluting Stents
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1-2010-0007
Record Dates: First submitted 2011-12-29; First posted 2012-01-02 (Estimated); Last update posted 2016-07-27 (Estimated); Status verified 2016-07

CONDITIONS: Stable Angina or Acute Coronary Syndrome Considered for Percutaneous Coronary Intervention With Dyslipidemia or Hypertension
Keywords: SES vs BES
MeSH Terms: conditions — Angina, Stable; Hypertension | interventions — Pravastatin; pitavastatin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (6):
- Cypher group (Active Comparator)
  Interventions: Device: Sirolimus-eluting stent
- Nobori group (Experimental)
  Interventions: Device: Biolimus-eluting stents
- Pravastatin group (Active Comparator)
  Interventions: Drug: pravastatin 20mg/day after DES implantation
- Pitivastatin group (Active Comparator)
  Interventions: Drug: pitavastatin 2mg/day after DES implantation
- Non-ARB group (Active Comparator)
  Interventions: Drug: Non-ARB /day after DES implantation
- ARB group (Experimental)
  Interventions: Drug: Eposartan 600mg/day after DES implantation

INTERVENTIONS:
Device: Sirolimus-eluting stent — 2x2 randomization by the treatment of dyslipidemia and hypertension(In patients of dyslipidemia: pitavastatin 2mg/day vs. pravastatin 20mg/day, in patients of hypertension: eporsartan 600mg/day vs. Non-ARB) and the types of the implanted DES, SES vs BES.
  Arms: Cypher group
Device: Biolimus-eluting stents — 2x2 randomization by the treatment of dyslipidemia and hypertension(In patients of dyslipidemia: pitavastatin 2mg/day vs. pravastatin 20mg/day, in patients of hypertension: eporsartan 600mg/day vs. Non-ARB) and the types of the implanted DES, SES vs BES.
  Arms: Nobori group
Drug: pravastatin 20mg/day after DES implantation — 2x2 randomization by the treatment of dyslipidemia and hypertension(In patients of dyslipidemia: pitavastatin 2mg/day vs. pravastatin 20mg/day, in patients of hypertension: eporsartan 600mg/day vs. Non-ARB) and the types of the implanted DES, SES vs BES.
  Arms: Pravastatin group
Drug: pitavastatin 2mg/day after DES implantation — 2x2 randomization by the treatment of dyslipidemia and hypertension(In patients of dyslipidemia: pitavastatin 2mg/day vs. pravastatin 20mg/day, in patients of hypertension: eporsartan 600mg/day vs. Non-ARB) and the types of the implanted DES, SES vs BES.
  Arms: Pitivastatin group
Drug: Non-ARB /day after DES implantation — 2x2 randomization by the treatment of dyslipidemia and hypertension(In patients of dyslipidemia: pitavastatin 2mg/day vs. pravastatin 20mg/day, in patients of hypertension: eporsartan 600mg/day vs. Non-ARB) and the types of the implanted DES, SES vs BES.
  Arms: Non-ARB group
Drug: Eposartan 600mg/day after DES implantation — 2x2 randomization by the treatment of dyslipidemia and hypertension(In patients of dyslipidemia: pitavastatin 2mg/day vs. pravastatin 20mg/day, in patients of hypertension: eporsartan 600mg/day vs. Non-ARB) and the types of the implanted DES, SES vs BES.
  Arms: ARB group

SUMMARY:
There has been little research on neointimal coverage and malapposition after BES implantation using OCT in human coronary artery. Furthermore, specific drug may possibly influence the vascular healing after stent implantation. Therefore, this study will investigate 1) neointimal coverage and malapposition on OCT after BES versus SES implantation and 2) relationship of specific drug treatment and neointimal coverage or late malapposition by the prospective, randomized study.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 20 year old
2. In the case that the blood pressure at rest is greater than systolic 140mmHg or more than diastolic 90mmHg
3. When someone is taking Anti-Hypertensive medication
4. If total cholesterol is more than 200mg/dL and LDL-cholesterol is greater than 130mg/dL or if you are taking a statin
5. Significant coronary de novo lesion (> 70% by quantitative angiographic analysis)
6. Patients with stable angina or acute coronary syndrome considered for percutaneous coronary intervention.
7. Reference vessel diameter of 2.5 to 3.5 mm by operator assessment
8. Stent size of 2.5 to 3.5 mm and stent length ≤ 24 mm

Exclusion Criteria:

1. Contraindication to anti-platelet agents
2. Proximal leison within 15 mm from ostium
3. Creatinine level 2.0 mg/dL or end stage renal disease on dialysis
4. Pregnant women or women with potential childbearing
5. Life expectancy less than 1 year
6. Complex lesion morphologies (aorto-ostial, bifurcation with >2.0 mm side branch, unprotected Left main, thrombus, severe calcification, chronic total occlusion)
7. Vein graft lesion

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2010-07; Primary Completion 2015-05 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
neointimal coverage | 6month
  1. To compare the neointimal coverage on 6-month follow-up OCT according to specific drug treatment in 2 patient subgroups at 6-month after DES implantation.
  2. To compare the neointimal coverage on 6-month follow-up OCT according to the randomly assigned BES or SES implantation.

SECONDARY OUTCOMES:
stent malapposition and thrombus | 6month
  The secondary endpoint of this study is to compare percent of stent malapposition and thrombus at 6 months according to specific drug treatment in 2 patient subgroups or to the types of implanted DES, SES vs. BES by a 6-month follow-up OCT.

CONTACTS AND LOCATIONS:
Overall Officials: Myeong Ki Hong, Ph.D, Principal Investigator — Severance Hospital
Locations (1):
- Severance Hospital, Seoul, Seoul, South Korea

REFERENCES:
- [Derived] Kim JS, Ha J, Kim BK, Shin DH, Ko YG, Choi D, Jang Y, Hong MK. The relationship between post-stent strut apposition and follow-up strut coverage assessed by a contour plot optical coherence tomography analysis. JACC Cardiovasc Interv. 2014 Jun;7(6):641-51. doi: 10.1016/j.jcin.2013.12.205. Epub 2014 May 14. PMID 24835329
- [Derived] Kim BK, Ha J, Mintz GS, Kim JS, Shin DH, Ko YG, Choi D, Jang Y, Hong MK. Randomised comparison of strut coverage between Nobori biolimus-eluting and sirolimus-eluting stents: an optical coherence tomography analysis. EuroIntervention. 2014;9(12):1389-97. doi: 10.4244/EIJV9I12A236. PMID 24531309